CLINICAL TRIAL: NCT07114926
Title: Study on the Function of Taiwan Green Propolis in Reducing Blood Lipids and Body Fat in Sub-healthy Groups: MASLD
Acronym: TGP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kuo,HSIN-YU (Other)
Responsible Party: Sponsor-Investigator, Kuo,HSIN-YU, Principal Investigator, Taipei Medical University
Organization: Taipei Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A11303004; A11303004 (Other Grant/Funding Number: Buddhist Tzu Chi Medical Foundation Dalin Tzu Chi Hospital); N202305017 (Other Grant/Funding Number: TMU-Joint Institutional Review Board)
Record Dates: First submitted 2025-07-01; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-07

CONDITIONS: MASLD - Metabolic Dysfunction-Associated Steatotic Liver Disease
Keywords: Taiwanese green propolis; MASLD-Metabolic Dysfunction-Associated Steatotic Liver Disease; blood lipids; body fat; Health Belief Model; quality of life

STUDY DESIGN:
Intervention Model Description: The study design adopted a parallel, double-blind, randomized approach to the experimental group (propolis) and the control group (placebo).
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Take two capsules of Taiwan Green Propolis (each containing 500 mg/mL of propolis) before breakfast and dinner daily, totaling four capsules/day for 12 consecutive weeks.
  Interventions: Dietary Supplement: Taiwanese green propolis
- Control group (Placebo Comparator): Take placebo capsules identical in appearance, smell, and content, with the same dosage and frequency.
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: Taiwanese green propolis — Intervention Details:
  Experimental Group: Take two capsules of Taiwan Green Propolis (each containing 500 mg/mL of propolis) before breakfast and dinner daily, totaling four capsules/day for 12 consecutive weeks.
  During the intervention period, both groups will maintain their usual diet and activity levels and receive the same health education on nutrition and exercise.
  Other Names: placebo
  Arms: Experimental Group
Dietary Supplement: placebo — Take placebo capsules identical in appearance, smell, and content, with the same dosage and frequency.
  Arms: Control group

SUMMARY:
This study investigates the effectiveness of Taiwanese green propolis in reducing blood lipids and body fat in sub-healthy individuals. The study design follows a parallel, double-blind, randomized assignment approach, dividing participants into an experimental group (propolis) and a control group (placebo). Researchers explained the study plan to participants, and after obtaining signed informed consent, participants were randomly assigned using a web-based program that generated random serial numbers. The randomization was stratified by gender (male-to-female ratio of 1:1) and physiological age groups (maturity, middle age, menopause, post-menopause, and old age). Serial numbers and group assignments were sequentially encoded and placed in opaque, consecutively numbered envelopes. After obtaining consent, researchers opened the sealed envelopes in order and assigned participants to either the experimental group (propolis) or the control group (placebo), with 30 participants in each group.

The experimental group received Taiwanese green propolis (which can be stored at room temperature) in capsule form, containing 500 mg/ml of propolis extract per capsule. Participants took two capsules before breakfast and two before dinner, totaling four capsules per day for 12 weeks. The control group received a placebo with the same dosage and administration method. All participants were instructed not to deliberately change their daily diet or exercise routines during the study. To assess adherence, participants recorded their daily propolis capsule intake. Additionally, the Health Belief Model questionnaire and the EQ-5D-5L quality of life questionnaire were used to evaluate whether the intervention with propolis, along with dietary and exercise education, contributed to increased awareness of health behaviors and improvements in quality of life.

The primary outcomes of the study include changes in blood lipids, body fat, blood glucose levels, liver fat, and liver fibrosis. The secondary outcomes focus on the correlation between health behavior awareness and quality of life.

Keywords: Taiwanese green propolis, sub-health, blood lipids, body fat, Health Belief Model, quality of life.

DETAILED DESCRIPTION:
Inclusion and Exclusion Criteria

Inclusion Criteria:

Aged 18 to 80 years.

Meet any of the following dyslipidemia indicators:

Total cholesterol (TC) > 200 mg/dL

Triglycerides (TG) > 200 mg/dL

LDL cholesterol > 130 mg/dL

Overweight or obese (BMI ≥ 27) with abnormal waist circumference:

Male > 90 cm

Female > 80 cm

Not currently receiving any lipid-lowering medication treatment.

Exclusion Criteria:

Allergic to honey, propolis, various pollens, or alcohol.

Individuals with psychiatric disorders or cognitive impairments.

Pregnant or breastfeeding women.

Individuals with significant endocrine disorders or major diseases of the heart, liver, kidneys, or other organs.

Individuals with swallowing difficulties.

Individuals with dementia, impaired consciousness, or other cognitive disorders preventing informed consent.

Individuals already receiving formal lipid-lowering drug therapy.

Individuals with comorbid diabetes, chronic kidney disease, or isolated LDL > 190 mg/dL.

ELIGIBILITY:
Inclusion Criteria:

Aged 18 to 80 years.

Meet any of the following dyslipidemia indicators:

Total cholesterol (TC) > 200 mg/dL

Triglycerides (TG) > 200 mg/dL

LDL cholesterol > 130 mg/dL

Overweight or obese (BMI ≥ 27) with abnormal waist circumference:

Male > 90 cm

Female > 80 cm

Not currently receiving any lipid-lowering medication treatment. MASLD

Exclusion Criteria:

* Allergic to honey, propolis, various pollens, or alcohol.

Individuals with psychiatric disorders or cognitive impairments.

Pregnant or breastfeeding women.

Individuals with significant endocrine disorders or major diseases of the heart, liver, kidneys, or other organs.

Individuals with swallowing difficulties.

Individuals with dementia, impaired consciousness, or other cognitive disorders preventing informed consent.

Individuals already receiving formal lipid-lowering drug therapy.

Individuals with comorbid diabetes, chronic kidney disease, or isolated LDL > 190 mg/dL.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08-30 (Estimated); Primary Completion 2028-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
In body | Time Points for Data Collection: Baseline (before intervention) Week 4, Week 8, and Week 12 of the intervention Follow-up at Week 2 and Week 12 after the intervention ends
  body fat composition
Changes in blood lipids | Baseline (before intervention) Week 4, Week 8, and Week 12 of the intervention Follow-up at Week 2 and Week 12 after the intervention ends
  TG, TC, HDL, LDL
fatty liver status | Time Points for Data Collection: Baseline (before intervention) Week 4, Week 8, and Week 12 of the intervention Follow-up at Week 2 and Week 12 after the intervention ends
  assessed via abdominal ultrasound

SECONDARY OUTCOMES:
Eating Behavior Scale | Time Points for Data Collection: Baseline (before intervention) Week 4, Week 8, and Week 12 of the intervention Follow-up at Week 2 and Week 12 after the intervention ends
  diet
quality of life Questionnaire Assessments | Time Points for Data Collection: Baseline (before intervention) Week 4, Week 8, and Week 12 of the intervention Follow-up at Week 2 and Week 12 after the intervention ends
  EQ-5D-5L Quality of Life Questionnaire The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state
gut microbiota | Collected at baseline and Week 12 to assess gut microbiota changes
  Stool Samples After collecting fecal samples, they are sent to Microbacteria Ark Company for testing of microbes at low temperature.
inflammatory markers | Baseline (before intervention) Week 4, Week 8, and Week 12 of the intervention Follow-up at Week 2 and Week 12 after the intervention ends
  (IL-6, IL-8, IL-1β)
health beliefs | Time Points for Data Collection: Baseline (before intervention) Week 4, Week 8, and Week 12 of the intervention Follow-up at Week 2 and Week 12 after the intervention ends
  Health Belief Questionnaire
ESAS Fatigue Scale | Time Points for Data Collection: Baseline (before intervention) Week 4, Week 8, and Week 12 of the intervention Follow-up at Week 2 and Week 12 after the intervention ends
  fatigue symptoms Please circle the number that best describes how you feel NOW Pain、 Tiredness、Drowsiness、Nausea、Lack of Appetitie、 Shortness of Breath、 Depression、Anxiety、Wellbeing 0 to 10 points, the lower the better
IPAQ | Baseline (bWeek 4, Week 8, and Week 12 of the intervention Follow-up at Week 2 and Week 12 after the intervention ends efore intervention)
  physical activity

CONTACTS AND LOCATIONS:
Locations (1):
- Buddhist Tzu Chi Medical Foundation Dalin Tzu Chi Hospital, Chiayi City, Dalin, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Collect all to IPD
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 2 years after publication
Access Criteria: 2 years after publication
URL: https://ohr.tmu.edu.tw/zh-Hant/news/375